CLINICAL TRIAL: NCT04883242
Title: Isa-CAPED MM: Isatuximab, Carfilzomib, Pomalidomide, and Dexamethasone (Isa-KPd) for Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Isatuximab, Carfilzomib, Pomalidomide, and Dexamethasone for the Treatment of Relapsed or Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1121154; NCI-2021-03406 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10690 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; isatuximab; pomalidomide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (isatuximab, carfilzomib, pomalidomide, steroid) (Experimental): INDUCTION: Patients receive isatuximab IV on days 1, 8, 15, and 22 of cycle 1 and days 1 and 15 of subsequent cycles carfilzomib IV over 30 minutes on days 1, 8, and 15, pomalidomide PO QD on days 1-21, and dexamethasone PO or IV on days 1,8, 15, and 22. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive isatuximab IV days 1 and 15, carfilzomib IV over 30 minutes on days 1 and 15, pomalidomide PO QD on days 1-21, and dexamethasone PO or IV on days 1, 8, 15, and 22. Cycles repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  All patients undergo bone marrow aspirate and biopsy during screening, skeletal x-ray, CT, PET-CT, or MRI, bone marrow and blood sample collection throughout the study.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Biological: Isatuximab; Drug: Pomalidomide; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration; Procedure: Skeletal Survey X-Ray; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Carfilzomib — Given IV
  Other Names: Kyprolis; PR-171; Carfilnat; CFZ
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Biological: Isatuximab — Given IV
  Other Names: Hu 38SB19; Isatuximab-irfc; SAR 650984; SAR650984; Sarclisa; SAR-650984
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Imnovid; Pomalyst; CC4047
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Skeletal Survey X-Ray — Undergo skeletal x-ray
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT Scan; Computed Axial Tomography
Procedure: Positron Emission Tomography — Undergo PET-CT
  Other Names: PET scan
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI

SUMMARY:
This phase II trial studies the effect of isatuximab, carfilzomib, pomalidomide, and dexamethasone in treating patients with multiple myeloma that has come back (relapsed) or does not respond to treatment (refractory). Isatuximab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Carfilzomib may stop the growth of cancer cells by blocking some of the proteins needed for cell growth. Pomalidomide may help shrink or slow the growth of multiple myeloma. Anti-inflammatory drugs, such as dexamethasone lower the body's immune response and are used with other drugs in the treatment of some types of cancer. Giving isatuximab, carfilzomib, pomalidomide, and dexamethasone may kill more cancer cells.

DETAILED DESCRIPTION:
OUTLINE:

INDUCTION: Patients receive isatuximab intravenously (IV) on days 1, 8, 15, and 22 of cycle 1 and days 1 and 15 of subsequent cycles carfilzomib IV over 30 minutes on days 1, 8, and 15, pomalidomide orally (PO) once daily (QD) on days 1-21, and dexamethasone PO or IV on days 1,8, 15, and 22. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive isatuximab IV days 1 and 15, carfilzomib IV over 30 minutes on days 1 and 15, pomalidomide PO QD on days 1-21, and dexamethasone PO or IV on days 1, 8, 15, and 22. Cycles repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

All patients undergo bone marrow aspirate and biopsy during screening, skeletal x-ray, computed tomography (CT), positron emission tomography (PET)-CT, or magnetic resonance imaging (MRI), bone marrow and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days, then for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory multiple myeloma, with >= 1 prior therapy
* Must have received prior lenalidomide therapy
* Must have measurable disease, as defined by International Myeloma Working Group criteria, having one or more of the following:

  * Serum M protein >= 0.5 g/dL
  * Urine M protein >= 200 mg/24 hours
  * Involved serum free light chain level >= 10 mg/dL with abnormal kappa/lambda ratio
  * Measurable biopsy-proven plasmacytomas (>= 1 lesion has a single diameter >= 2 cm)
  * Bone marrow plasma cells >= 30%
* Age 18 years and older, and have the capacity to give informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Subjects should have resolution of any toxicities from prior therapy to grade =< 1 or baseline prior to enrollment (with the exception of peripheral neuropathy)
* Subjects are required to have grade =< 2 peripheral neuropathy to enroll
* Prior autologous stem cell transplant is allowed; patients must be >= 6 months post- autologous stem cell transplantation to enroll
* Estimated glomerular filtration rate (eGFR) >= 20 ml/min
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN)
* Total bilirubin =< 2 x ULN
* Absolute neutrophil count (ANC) >= 1,000/uL
* Platelets >= 50,000/uL
* Hemoglobin >= 8 g/dL
* Growth factor use or transfusions may be used to meet the eligibility requirement for ANC, platelets, and hemoglobin
* Female patients of childbearing potential and male patients must agree to use 2 effective forms of contraception or continuously abstain from heterosexual intercourse during the period of therapy, and for 6 months after discontinuation of study treatment for females and 3 months after discontinuation of study treatment for males

Exclusion Criteria:

* History of clinically significant cardiovascular disease, including congestive heart failure New York Heart Association (NYHA) class 3-4, symptomatic ischemia, left ventricular ejection fraction < 40%, uncontrolled conduction abnormalities, myocardial infarction in last 6 months
* Uncontrolled hypertension as determined by the principal investigator (PI) or designee
* Active plasma cell leukemia or systemic amyloid light-chain (AL) amyloidosis
* History of another primary malignancy that has not been in remission for at least 1 year

  * However, the following diagnoses are eligible for inclusion: non-melanoma skin cancer, localized prostate cancer, superficial bladder cancer, cervical carcinoma in situ, on biopsy or any prior malignancy with an estimated > 90% 1-year cure rate per sponsor-investigator
* For patients with chronic hepatitis B viral infection, the hepatitis B virus (HBV) polymerase chain reaction (PCR) must be undetectable on suppressive therapy
* Patients with a history of Hepatitis C viral infection must have been treated and cured. For patients on treatment for hepatitis C, they are eligible if they have an undetectable hepatitis C virus (HCV) viral load
* Subjects with active uncontrolled infection
* Concurrent use of other anticancer agents or experimental treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to 5 years post treatment
  Responses will be based on the International Myeloma Working Group criteria for response in multiple myeloma.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From first study drug administration to the first occurrence of disease progression or death from any cause, assessed up to 5 years
  PFS will be calculated using assessments by investigators. Kaplan-Meier methodology will be used to estimate event-free curves and corresponding quartiles (including the median).
Overall survival | From the first study drug administration to death from any cause, assessed up to 5 years
  Kaplan-Meier methodology will be used to estimate the event-free curves.
Duration of response | Up to 5 years post treatment
Time to progression | Up to 5 years post treatment
Incidence of adverse events | Up to 30 days post treatment
  Will be measured by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Rates of minimal residual disease negativity | Up to 5 years post treatment
  Measured by next-generation sequencing of immunoglobulin genes in the bone marrow.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Banerjee, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT04883242/ICF_000.pdf